CLINICAL TRIAL: NCT01330927
Title: A Randomised, Double-blind, Placebo-controlled, Five-way Cross-over Dose Response Study to Determine the Effect of VA106483 on Nocturnal Urine Volume in Elderly Male Subjects With Nocturia and Benign Prostatic Hypertrophy (BPH)
Brief Title: Dose Response Study of VA106483 in Males With Nocturia and Benign Prostatic Hypertrophy (BPH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Dr Hilary McElwaine-Johnn / Chief Medical Officer, Vantia Ltd, 1 Venture Road, Southampton Science Park, Southampton, SO16 7NP, UK
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 483-008
Record Dates: First submitted 2011-03-30; First posted 2011-04-07 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Nocturia; Benign Prostatic Hypertrophy (BPH)
Keywords: VA106483; Nocturia; Benign Prostatic Hypertrophy; BPH; Elderly; Males; Nocturnal voids; Anti-diuretic
MeSH Terms: conditions — Nocturia; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- VA106483 0.5 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 1 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 2 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 4 mg (Experimental)
  Interventions: Drug: VA106483
- Sugar pill (Placebo Comparator)
  Interventions: Drug: VA106483

INTERVENTIONS:
Drug: VA106483 — Once daily oral dose of placebo for 2 nights
  Once daily oral dose of 0.5 mg VA106483 for 2 nights
  Once daily oral dose of 1 mg VA106483 for 2 nights
  Once daily oral dose of 2 mg VA106483 for 2 nights
  Once daily oral dose of 4 mg VA106483 for 2 nights
  Placebo: as above

SUMMARY:
The purpose of this study is to establish the dose response relationship of VA106483 and nocturnal urine volumes in a population of elderly male subjects with Benign Prostatic Hypertrophy (BPH) who are likely to present with nocturia.

DETAILED DESCRIPTION:
VA106483 is a selective vasopressin V2-receptor (V2-receptor) agonist that is being developed for the treatment of nocturia.

The antidiuretic effect of V2-receptor stimulation in the kidneys is well established through the use of the peptide agonist, desmopressin, which shows clinical benefit in diabetes insipidus, primary nocturnal enuresis and nocturia.

Nocturia, defined as waking to void at least once per night between periods of sleep, is a common complaint and shows an age-dependent increase in both prevalence and severity (number of nocturnal voids). It is the most bothersome symptom of benign prostatic hypertrophy and has been linked to an age-dependent loss in circadian release of endogenous nocturnal vasopressin and consequent over production of urine at night (nocturnal polyuria).

Correlation between nocturnal urine volume and nocturnal void frequency has been demonstrated in previous studies of V2-receptor agonists.

The purpose of this study is to determine the dose response relationship of VA106483 and nocturnal urine volumes.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 65 years old and above with history of nocturia and benign prostatic hypertrophy (BPH)

Exclusion Criteria:

* Administration of any Investigational Medicinal Product (IMP) within 10 weeks before entry to the study
* Any clinically significant concomitant medical disease, condition or abnormal laboratory test result
* Other protocol defined eligibility criteria may apply

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in the mean nocturnal urine volumes | 20 days

SECONDARY OUTCOMES:
Change in the mean nocturnal void frequency | 20 days
Change in mean time to first void | 20 days
Change in frequency of daytime voids | 20 days
Change in mean volume of daytime voids | 20 days
Change in mean nocturnal urine osmolality | 20 days
Change in mean daytime urine osmolality | 20 days
Change in mean voided volumes | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Georg Golor, PD Dr. med., Principal Investigator — Parexel
Locations (1):
- Early Phase Clinical Unit, PAREXEL International GmbH, Berlin, Germany